CLINICAL TRIAL: NCT05114902
Title: Assessing the Impact of PCV13 on Pneumococcal Nasopharyngeal Colonization in Children 8 Weeks to ≤60 Months of Age Hospitalized for Pneumonia in the Philippines
Brief Title: PCV13 Impact on Pneumococcal Nasopharyngeal Carriage Study
Acronym: IMPACT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Asian Foundation for Tropical Medicine Inc. (Other)
Collaborators: Pfizer (Industry); Philippine Children's Medical Center, Philippines (Unknown); Southern Philippines Medical Center (Other)
Responsible Party: Principal Investigator, Marilla Lucero, Principal Investigator, Asian Foundation for Tropical Medicine Inc.
Other Study IDs: CT-44 Study Protocol AFTM-01
Record Dates: First submitted 2021-10-29; First posted 2021-11-10 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Community-acquired Pneumonia
Keywords: Clinical CAP
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The retained specimen will consist of isolates of Streptococcus pneumoniae cultured from the nasopharyngeal swab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PCV13 Non-vaccinated Settting: Pneumococcal vaccine-naïve children at the PCMC
  Interventions: Diagnostic Test: Nasopharyngeal swab
- PCV13 Vaccinated Setting: Pneumococcal vaccine-exposed children at the SPMC
  Interventions: Diagnostic Test: Nasopharyngeal swab

INTERVENTIONS:
Diagnostic Test: Nasopharyngeal swab — A sample obtained from the nasopharynx for detection of live pneumococci and pneumococcal respiratory carriage

SUMMARY:
Prospective, observational, hospital based, nasopharyngeal carriage (NPC), vaccine effectiveness study Comparisons will be made in Filipino children, aged 8 weeks to ≤60 months of age at enrollment, who have been hospitalized with a radiologically-confirmed, community-acquired pneumonia (CAP).

DETAILED DESCRIPTION:
This study will be the first of two phases (A and B). Phase A will compare a PCV13-vaccinated setting (SPMC) with an unvaccinated setting (PCMC)

ELIGIBILITY:
Inclusion Criteria:

1. Child 8 weeks to ≤60 months of age
2. Resident of the National Capital Region (NCR) or Region X-XIII
3. Child admitted with a medical diagnosis of clinical CAP based on history and physical exam
4. Written informed consent obtained from a parent or legal guardian
5. At SPMC site, child must have received at least 1 dose of PCV13 given at <12 months based on history-taking
6. For Phase B at PCMC site, child must have received at least 1 dose of PCV13 given at <12 months based on history-taking

Exclusion Criteria:

1. Children with a known primary or secondary immunodeficiency
2. Child with a contraindication to doing a nasopharyngeal swab which may include, but is not limited to: dyscrasias, coagulation disorders, or other diseases (e.g., hemophilia, purpura), presence of craniofacial abnormalities32
3. For Phase A at PCMC site, child with any PCV in the past based on history-taking

Ages: 8 Weeks to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children 8 weeks to ≤60 months of age from the National Capital Region (NCR) or Region X-XIII admitted with a medical diagnosis of clinical community-acquired pneumonia (CAP), confirmed by an abnormal chest x-ray. In Region X-XIII, the child must have received at least 1 dose of PCV13 given at <12 months.
Sampling Method: Non-Probability Sample
Enrollment: 451 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
S. pneumoniae serotypes | Upon Admission
  S. pneumonia serotypes isolated from the nasopharynx of children admitted in PCV13-unvaccinated site (PCMC)
S. pneumoniae serotypes Upon Admission | Upon Admission
  S. pneumonia serotypes isolated from the nasopharynx of children admitted in PCV13-unvaccinated site (SPMC)
Antimicrobial resistance rate of S. pneumoniae | Upon Admission
  Antimicrobial resistance rate isolated from the nasopharynx of children admitted as a case of radiologic CAP admitted in PCV13- unvaccinated site (PCMC)
Antimicrobial resistance rate of S. pneumoniae | Upon Admission
  Antimicrobial resistance rate isolated from the nasopharynx of children admitted as a case of radiologic CAP admitted in PCV13-vaccinated site (SPMC)

CONTACTS AND LOCATIONS:
Overall Officials: Marilla G Lucero, MD, Principal Investigator — Asian Foundation for Tropical Medicine
Locations (1):
- Philippine Children's Medical Center, Quezon City, National Capital Region, Philippines